CLINICAL TRIAL: NCT05507476
Title: Effects of Nasal Desmopressin Spray Versus Topical Epinephrine on Surgical Field Clarity and Hemodynamics in Endonasal Dacryocystorhinostomy: a Randomized Clinical Study.
Brief Title: Nasal Desmopressin Versus Topical Epinephrine in Endonasal Dacryocystorhinostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Nasal Desmopressin in DCR
Record Dates: First submitted 2022-08-14; First posted 2022-08-19 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2023-06

CONDITIONS: Anesthesia
Keywords: Desmopressin; Dacryocystorhinostomy
MeSH Terms: interventions — Deamino Arginine Vasopressin; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Desmopressin group (Active Comparator): The patient will receive two puffs of desmopressin acetate 10 µg/puff in the side of the nasal cavity ipsilateral to the obstructed lacrimal duct (20 μg totally) 60 minutes before surgery "Minirin 10 μg/0.1 ml per spray, Ferring Pharmaceutical Company". Three normal saline-soaked packs will be placed in the middle meatus for 5 minutes immediately before the start of surgery.
  Interventions: Drug: Desmopressin Acetate Nasal, 10 μg/0.1 ml per spray
- Epinephrine group (Active Comparator): The patient will receive topical 1:100,000 epinephrine in the side of the nasal cavity ipsilateral to the obstructed lacrimal duct via 3 soaked packs placed in the middle meatus for 5 minutes immediately before the start of surgery. The patient will also receive two puffs of normal saline "prepared in emptied Minirin bottle" in the same nasal cavity 60 minutes before surgery.
  Interventions: Drug: Epinephrine topical 1:100,000 Nasal Packs

INTERVENTIONS:
Drug: Desmopressin Acetate Nasal, 10 μg/0.1 ml per spray — The patient will receive two puffs of desmopressin acetate 10 µg/puff in the side of the nasal cavity ipsilateral to the obstructed lacrimal duct (20 μg totally) 60 minutes before surgery.
  Other Names: Minirin 10 μg/0.1 ml per spray
  Arms: Desmopressin group
Drug: Epinephrine topical 1:100,000 Nasal Packs — The patient will receive topical 1:100,000 epinephrine in the side of the nasal cavity ipsilateral to the obstructed lacrimal gland via 3 soaked packs placed in the middle meatus for 5 minutes immediately before the start of surgery.
  Other Names: Adrenaline 1 mg / 1ml
  Arms: Epinephrine group

SUMMARY:
Dacryocystorhinostomy aims to create a channel between the lacrimal sac and nasal mucosa to relieve nasolacrimal duct occlusion. General anesthesia is still preferred by many surgeons to secure the airway and control blood pressure.

DETAILED DESCRIPTION:
Bleeding even minor can obscure the surgical field. This can extend the operative time & increase the failure rate. The hemostatic effect of desmopressin on the quality of the surgical field was investigated in patients undergoing endoscopic sinus surgery and revealed that desmopressin could reduce intraoperative bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-45 years old.
* Physical status: ASA I & II.
* Type of operations: elective endonasal dacryocystorhinostomy under general anesthesia.
* Written informed consent from the patient.

Exclusion Criteria:

* Patient refusal.
* Known hypersensitivity to study drugs.
* Nasal pathology as active infection or an anatomical abnormality.
* Hyponatremia "serum Na+ less than 135".
* Coagulation disorders.
* Renal or cardiovascular disorders.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss | Measurement will be done at the 30th minutes of the start of surgery.
  Estimation of intraoperative blood loss will be done at 30th minutes of surgery.
  by calculating the loss of blood and irrigation saline in 50 mL-graded suction canisters.
Intraoperative blood loss | Measurement will be done at 60th minutes of the start of surgery.
  Estimation of intraoperative blood loss will be done at 60th minutes of surgery.
  by calculating the loss of blood and irrigation saline in 50 mL-graded suction canisters.

SECONDARY OUTCOMES:
The Surgical field clarity | at the end of surgery
  The quality of surgical field based on BOEZAART grading system(0 no bleeding; 1 slight bleeding: no suctioning is needed; 2 slight bleeding: occasional suctioning needed;, 3 sight bleeding: frequent suctioning required, bleeding threatens surgical field a few seconds after suction is removed; 4 moderate bleeding: frequent suctioning required and bleeding threatens surgical field directly after suction is removed; 5 severe bleeding: constant suctioning required)
Change in heart rate (HR) in beat per minute | will be recorded at 2 minutes, 5 minutes, 10 minutes, 30 minutes and 60 minutes after topical epinephrine packs insertion.
  Change in heart rate (HR) from baseline.
Change mean arterial blood pressure (MAP) in mmHg | will be recorded at 2 minutes, 5 minutes, 10 minutes, 30 minutes and 60 minutes after topical epinephrine packs insertion.
  Change mean arterial blood pressure (MAP) from baseline.
Change oxygen saturation (SPO2) | will be recorded at 2 minutes, 5 minutes, 10 minutes, 30 minutes and 60 minutes after topical epinephrine packs insertion.
  Change oxygen saturation (SPO2) from baseline.
Change in serum sodium level | preoperative and after 12 hours postoperative
  Serum sodium level will be measured pre & postoperative to detect and manage any sodium disturbances.
The surgeon's satisfaction | At the end of surgery
  The surgeon was asked to rate satisfaction at the end of surgery (4 =excellent, 3 = good, 2 = fair, 1 = poor, 0 = extremely poor).

CONTACTS AND LOCATIONS:
Overall Officials: Alshaimaa Abdel Fattah Kamel, MD, Principal Investigator — Assistant professor of Anesthesia, Intensive Care & Pain management,Zagazig University; Marwa Ahmed Mohamed Khedr, MD, Principal Investigator — Lecturer of Ophthalmology, Zagazig University
Locations (1):
- Zagazig university hospital, Zagazig, Al-Sharkia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vinciguerra A, Nonis A, Giordano Resti A, Ali MJ, Bussi M, Trimarchi M. Role of anaesthesia in endoscopic and external dacryocystorhinostomy: A meta-analysis of 3282 cases. Eur J Ophthalmol. 2022 Jan;32(1):66-74. doi: 10.1177/11206721211035616. Epub 2021 Jul 28. PMID 34318721
- [Background] Shao H, Kuang LT, Hou WJ, Zhang T. Effect of desmopressin administration on intraoperative blood loss and quality of the surgical field during functional endoscopic sinus surgery: a randomized, clinical trial. BMC Anesthesiol. 2015 Apr 17;15:53. doi: 10.1186/s12871-015-0034-8. PMID 25895497
- [Background] Jahanshahi J, Tayebi E, Hashemian F, Bakhshaei MH, Ahmadi MS, Seif Rabiei MA. Effect of local desmopressin administration on intraoperative blood loss and quality of the surgical field during functional endoscopic sinus surgery in patients with chronic rhinosinusitis: a triple-blinded clinical trial. Eur Arch Otorhinolaryngol. 2019 Jul;276(7):1995-1999. doi: 10.1007/s00405-019-05435-3. Epub 2019 Jun 3. PMID 31161361
- [Background] Gruber RP, Zeidler KR, Berkowitz RL. Desmopressin as a hemostatic agent to provide a dry intraoperative field in rhinoplasty. Plast Reconstr Surg. 2015 May;135(5):1337-1340. doi: 10.1097/PRS.0000000000001158. PMID 25919247
- [Background] Korkmaz H, Yao WC, Korkmaz M, Bleier BS. Safety and efficacy of concentrated topical epinephrine use in endoscopic endonasal surgery. Int Forum Allergy Rhinol. 2015 Dec;5(12):1118-23. doi: 10.1002/alr.21590. Epub 2015 Jul 8. PMID 26152362
- [Background] Boezaart AP, van der Merwe J, Coetzee A. Comparison of sodium nitroprusside- and esmolol-induced controlled hypotension for functional endoscopic sinus surgery. Can J Anaesth. 1995 May;42(5 Pt 1):373-6. doi: 10.1007/BF03015479. PMID 7614641